CLINICAL TRIAL: NCT02775435
Title: A Randomized, Double-Blind, Phase III Study of Carboplatin-Paclitaxel/Nab-Paclitaxel Chemotherapy With or Without Pembrolizumab (MK-3475) in First Line Metastatic Squamous Non-small Cell Lung Cancer Subjects (KEYNOTE-407)
Brief Title: A Study of Carboplatin-Paclitaxel/Nab-Paclitaxel Chemotherapy With or Without Pembrolizumab (MK-3475) in Adults With First Line Metastatic Squamous Non-small Cell Lung Cancer (MK-3475-407/KEYNOTE-407)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-407; 173568 (Registry Identifier: JAPIC-CTI); MK-3475-407 (Other: MSD Protocol Number); KEYNOTE-407 (Other: MSD); 2016-000229-38 (EudraCT Number)
Record Dates: First submitted 2016-05-15; First posted 2016-05-17 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Chemotherapy Combo (Experimental): Participants receive pembrolizumab 200 mg by intravenous (IV) infusion prior to chemotherapy on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (~ 2 years) PLUS Investigator's choice of paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) or nab-paclitaxel (100 mg/m^2 by IV infusion on Days 1, 8, 15 of each 21-day cycle for 4 cycles) PLUS carboplatin area under the curve (AUC) 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Carboplatin
- Placebo + Chemotherapy (Active Comparator): Participants receive normal saline as placebo by IV infusion prior to chemotherapy on Day 1 of each 21-day cycle for up to 35 cycles (~ 2 years) PLUS Investigator's choice of paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) or nab-paclitaxel (100 mg/m^2 by IV infusion on Days 1, 8, 15 of each 21-day cycle for 4 cycles) PLUS carboplatin AUC 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
  Interventions: Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Saline placebo for pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Chemotherapy Combo
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®
Drug: Nab-paclitaxel — IV infusion
  Other Names: ABRAXANE®
Drug: Carboplatin — IV infusion Carboplatin dose should not to exceed 900 mg.
  Other Names: PARAPLATIN®
Drug: Saline placebo for pembrolizumab — IV infusion
  Arms: Placebo + Chemotherapy

SUMMARY:
This is a study of carboplatin and paclitaxel or nano particle albumin-bound paclitaxel (nab-paclitaxel) with or without pembrolizumab (MK-3475, KEYTRUDA®) in adults with first line metastatic squamous non-small cell lung cancer (NSCLC).

The primary hypotheses are that treatment with pembrolizumab prolongs: 1) Progression-free Survival (PFS) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by a blinded central imaging vendor compared to placebo, and 2) Overall Survival (OS).

After analysis of interim results was conducted, the protocol was amended (Amendment 5) to allow participants the option to discontinue placebo in the control arm and to switch to pembrolizumab in the event of documented progressive disease as assessed by central review.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of stage IV (M1a or M1b-American Joint Committee on Cancer [AJCC] 7th edition) squamous NSCLC.
* Has measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment.
* Has not received prior systemic treatment for metastatic NSCLC.
* Has provided tumor tissue from locations not radiated prior to biopsy.
* Has a life expectancy of at least 3 months.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Has adequate organ function.
* If female of childbearing potential, is willing to use an adequate method of contraception for the course of the study through 180 days after the last dose of study drug.
* If male with a female partner(s) of child-bearing potential, must agree to use an adequate method of contraception starting with the first dose of study drug through 95 days after the last dose of study drug. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

Exclusion Criteria:

* Has non-squamous histology NSCLC.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to administration of pembrolizumab.
* Before the first dose of study drug: a) Has received prior systemic cytotoxic chemotherapy for metastatic disease; b) Has received other targeted or biological antineoplastic therapy (e.g., erlotinib, crizotinib, cetuximab) for metastatic disease; c) Has had major surgery (<3 weeks prior to first dose).
* Received radiation therapy to the lung that is > 30 Gy within 6 months of the first dose of study drug.
* Completed palliative radiotherapy within 7 days of the first dose of study drug.
* Is expected to require any other form of antineoplastic therapy while on study.
* Has received a live-virus vaccination within 30 days of planned treatment start.
* Has a known history of prior malignancy except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has pre-existing peripheral neuropathy that is ≥ Grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) version 4 criteria.
* Previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Has a known sensitivity to any component of carboplatin or paclitaxel or nab-paclitaxel.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Is on chronic systemic steroids.
* Had prior treatment with any other anti-programmed cell death 1 (anti-PD-1), or programmed cell death ligand 1 (PD-L1) or PD-L2 agent or an antibody or a small molecule targeting other immuno-regulatory receptors or mechanisms.
* Has participated in any other pembrolizumab trial and has been treated with pembrolizumab.
* Has an active infection requiring therapy.
* Has known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or C. Active Hepatitis B.
* Is, at the time of providing documented informed consent, a regular user (including "recreational use") of any illicit drugs or has a recent history (within the last year) of substance abuse (including alcohol).
* Has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Garassino MC, Cheng Y, Rodriguez-Abreu D, Novello S, Mazieres J, Robinson AG, Powell SF, Halmos B, Gray JE, Wang M, Chen C, Yang J, Souza F, Schwarzenberger P, Paz-Ares L. Impact of Tumor Response and Response Duration on Survival Among Participants Receiving Pembrolizumab Plus Chemotherapy as First-Line Therapy for Non-Small-Cell Lung Cancer. Oncol Ther. 2025 Sep;13(3):667-681. doi: 10.1007/s40487-025-00350-6. Epub 2025 Jun 11. PMID 40498298
- [Derived] Cheng Y, Yang JC, Okamoto I, Zhang L, Hu J, Wang D, Hu C, Zhou J, Wu L, Cao L, Liu J, Zhang H, Sun H, Wang Z, Gao H, Yan Y, Xiao S, Lin J, Pietanza MC, Kurata T. Pembrolizumab plus chemotherapy for advanced non-small-cell lung cancer without tumor PD-L1 expression in Asia. Immunotherapy. 2023 Sep;15(13):1029-1044. doi: 10.2217/imt-2023-0043. Epub 2023 Jul 19. PMID 37465924
- [Derived] Garassino MC, Gadgeel S, Novello S, Halmos B, Felip E, Speranza G, Hui R, Garon EB, Horinouchi H, Sugawara S, Rodriguez-Abreu D, Reck M, Cristescu R, Aurora-Garg D, Loboda A, Lunceford J, Kobie J, Ayers M, Piperdi B, Pietanza MC, Paz-Ares L. Associations of Tissue Tumor Mutational Burden and Mutational Status With Clinical Outcomes With Pembrolizumab Plus Chemotherapy Versus Chemotherapy For Metastatic NSCLC. JTO Clin Res Rep. 2022 Nov 8;4(1):100431. doi: 10.1016/j.jtocrr.2022.100431. eCollection 2023 Jan. PMID 36793385
- [Derived] Novello S, Kowalski DM, Luft A, Gumus M, Vicente D, Mazieres J, Rodriguez-Cid J, Tafreshi A, Cheng Y, Lee KH, Golf A, Sugawara S, Robinson AG, Halmos B, Jensen E, Schwarzenberger P, Pietanza MC, Paz-Ares L. Pembrolizumab Plus Chemotherapy in Squamous Non-Small-Cell Lung Cancer: 5-Year Update of the Phase III KEYNOTE-407 Study. J Clin Oncol. 2023 Apr 10;41(11):1999-2006. doi: 10.1200/JCO.22.01990. Epub 2023 Feb 3. PMID 36735893
- [Derived] Paz-Ares L, Vicente D, Tafreshi A, Robinson A, Soto Parra H, Mazieres J, Hermes B, Cicin I, Medgyasszay B, Rodriguez-Cid J, Okamoto I, Lee S, Ramlau R, Vladimirov V, Cheng Y, Deng X, Zhang Y, Bas T, Piperdi B, Halmos B. A Randomized, Placebo-Controlled Trial of Pembrolizumab Plus Chemotherapy in Patients With Metastatic Squamous NSCLC: Protocol-Specified Final Analysis of KEYNOTE-407. J Thorac Oncol. 2020 Oct;15(10):1657-1669. doi: 10.1016/j.jtho.2020.06.015. Epub 2020 Jun 26. PMID 32599071
- [Derived] Mazieres J, Kowalski D, Luft A, Vicente D, Tafreshi A, Gumus M, Laktionov K, Hermes B, Cicin I, Rodriguez-Cid J, Wilson J, Kato T, Ramlau R, Novello S, Reddy S, Kopp HG, Piperdi B, Li X, Burke T, Paz-Ares L. Health-Related Quality of Life With Carboplatin-Paclitaxel or nab-Paclitaxel With or Without Pembrolizumab in Patients With Metastatic Squamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2020 Jan 20;38(3):271-280. doi: 10.1200/JCO.19.01348. Epub 2019 Nov 21. PMID 31751163
- [Derived] Paz-Ares L, Luft A, Vicente D, Tafreshi A, Gumus M, Mazieres J, Hermes B, Cay Senler F, Csoszi T, Fulop A, Rodriguez-Cid J, Wilson J, Sugawara S, Kato T, Lee KH, Cheng Y, Novello S, Halmos B, Li X, Lubiniecki GM, Piperdi B, Kowalski DM; KEYNOTE-407 Investigators. Pembrolizumab plus Chemotherapy for Squamous Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2040-2051. doi: 10.1056/NEJMoa1810865. Epub 2018 Sep 25. PMID 30280635
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26124&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response/progression, or adverse events during the second and switch-over pembrolizumab course were not counted towards efficacy outcome measures or safety outcome measures.
Groups:
- Pembrolizumab + Chemotherapy Combo: Participants received pembrolizumab 200 mg by intravenous (IV) infusion prior to chemotherapy on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (~ 2 years) PLUS Investigator's choice of paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) or nab-paclitaxel (100 mg/m^2 by IV infusion on Days 1, 8, 15 of each 21-day cycle for 4 cycles) PLUS carboplatin Area Under Curve (AUC) 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles. Participants who received pembrolizumab 200 mg IV Day 1 of 21-day cycle for up to 2 years, but experienced disease progression, were eligible to receive a second course of pembrolizumab 200 mg IV Day 1 of 21-day cycle, at the investigator's discretion, for 17 cycles (~ 1 year additional).
- Placebo + Chemotherapy: Participants received normal saline as placebo by IV infusion prior to chemotherapy on Day 1 of 21-day cycle for up to 35 cycles (~ 2 years) PLUS Investigator's choice of paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) or nab-paclitaxel (100 mg/m^2 by IV infusion on Days 1, 8, 15 of each 21-day cycle for 4 cycles) PLUS carboplatin AUC 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles. Participants with documented disease progression following placebo chemotherapy combo could switch-over to receive pembrolizumab for up to 35 cycles (~ 2 years). Eligible cross over participants who stopped pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (~ 1 year additional).
Period: Overall Study
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy
Started | 278 | 281
Treated | 278 | 280
Received Second Course of Pembrolizumab | 12 | 0
Received Switch-over Plus Second Course of Pembrolizuamb | 0 | 1
Switched to Pembrolizumab + Chemotherapy | 0 | 118
Completed | 0 | 0
Not Completed | 278 | 281
Not completed — Adverse Event | 32 | 27
Not completed — Lost to Follow-up | 2 | 2
Not completed — Sponsor decision | 44 | 19
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Death | 196 | 224

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy | Total
Number analyzed (Participants) | 278 | 281 | 559
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (8.8) | 64.8 (8.7) | 64.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 46 | 104
  Male | 220 | 235 | 455
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 56 | 52 | 108
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 4 | 7
  White | 216 | 214 | 430
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 9 | 11
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Expression Level: Tumor Proportion Score (TPS) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Participants with a TPS ≥1% were classified as PD-L1 positive and participants with a TPS <1% were classified as not PD-L1 positive.
  Participants
    TPS <1% | 95 | 99 | 194
    TPS ≥1% | 176 | 177 | 353
    Unknown | 7 | 5 | 12
Taxane Chemotherapy [Count of Participants; unit: Participants] — Participants were classified according to their taxane chemotherapy regimen: paclitaxel or nab-paclitaxel.
  Participants
    +Paclitaxel | 169 | 167 | 336
    +Nab-paclitaxel | 109 | 114 | 223
Geographic Region [Count of Participants; unit: Participants] — Participants were classified according to their geographic region: East Asia vs. non-East Asia.
  Participants
    East Asia | 54 | 52 | 106
    Non-East Asia | 224 | 229 | 453

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Criteria in Solid Tumors version 1.1 (RECIST 1.1), PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of ≥1 new lesions was also considered PD. PFS as assessed by blinded independent central review per RECIST 1.1 is presented.
Time Frame: Up to approximately 19 months
Population: The Intent-To-Treat population consisted of all randomized participants, regardless of whether or not they received study treatment. Participants were included in the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy
Number analyzed (Participants) | 278 | 281
Months | 6.4 [6.2 to 8.3] | 4.8 [4.3 to 5.7]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy Combo vs Placebo + Chemotherapy; Test type: Superiority; p < 0.0001, Regression, Cox — Treatment comparison stratified by programmed cell death-ligand 1 (PD-L1) status (Tumor Proportion Score [TPS] ≥1% vs. <1%), taxane chemotherapy (paclitaxel vs. nab-paclitaxel) & geographic region (East Asia vs. non-East Asia); Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.45 to 0.70]

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. OS is presented.
Time Frame: Up to approximately 19 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy
Number analyzed (Participants) | 278 | 281
Months | 15.9 [13.2 to NA] — NA=OS upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 11.3 [9.5 to 14.8]
Statistical Analysis 1: Comparison: Pembrolizumab + Chemotherapy Combo vs Placebo + Chemotherapy; Test type: Superiority; p = 0.0008, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.49 to 0.85]

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by RECIST 1.1. ORR as assessed by blinded independent central review per RECIST 1.1 is presented.
Time Frame: Up to approximately 19 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy
Number analyzed (Participants) | 278 | 281
Percentage of Participants | 57.9 [51.9 to 63.8] | 38.4 [32.7 to 44.4]

4. Secondary Outcome: Duration of Response (DOR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: For participants who demonstrated a confirmed response (Complete Response [CR]: Disappearance of all target lesions or Partial Response [PR]: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression as assessed by RECIST 1.1 or death. DOR as assessed by blinded independent central review per RECIST 1.1 is presented.
Time Frame: Up to approximately 19 months
Population: The Intent-To-Treat population consisted of all randomized participants, regardless of whether or not they received study treatment, who demonstrated a confirmed response (CR or PR). Participants were included in the treatment arm to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy
Number analyzed (Participants) | 161 | 108
Months | 7.7 [1.1 to 14.7] | 4.8 [1.3 to 15.8]

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 83 months
Population: The Safety population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy
Number analyzed (Participants) | 278 | 280
Participants | 274 | 275

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE was presented.
Time Frame: Up to approximately 29 months
Population: The Safety population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy
Number analyzed (Participants) | 278 | 280
Participants | 80 | 37

ADVERSE EVENTS:
Time Frame: Up to approximately 83 months
Description: All-Cause Mortality (ACM): all randomized participants. AEs: all participants who got ≥1 dose of study drug. Per protocol disease progression of cancer was not considered an AE unless related to study drug; MedDRA terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" unrelated to study drug are excluded as AEs. Per protocol, participants receiving switch-over, second course, and switch-over plus second course treatment were monitored for ACM and AEs separately.
Groups:
- Pembrolizumab + Chemotherapy Combo: Participants received pembrolizumab 200 mg by intravenous (IV) infusion prior to chemotherapy on Day 1 of 21-day cycle for up to 35 cycles PLUS Investigator's choice of paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) or nab paclitaxel (100 mg/m^2 by IV infusion on Days 1, 8, 15 of each 21-day cycle for 4 cycles) PLUS carboplatin Area Under Curve (AUC) 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
- Placebo + Chemotherapy: Participants received normal saline as placebo by IV infusion prior to chemotherapy on Day 1 of each 21-day cycle for up to 35 cycles (~ 2 years) PLUS Investigator's choice of paclitaxel (200 mg/m^2 by IV infusion on Day 1 of each 21-day cycle for 4 cycles) or nab-paclitaxel (100 mg/m^2 by IV infusion on Days 1, 8, 15 of each 21-day cycle for 4 cycles) PLUS carboplatin AUC 6 by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
- Placebo Switched Over to Pembrolizumab: Participants who received saline placebo with chemotherapy and who experienced disease progression, switched over to receive pembrolizumab monotherapy at investigator's discretion. Pembrolizumab was administered at 200 mg IV on Day 1 of each 21-day cycle for 35 cycles (~ 2 years).
- Pembrolizumab Combo (Second Course): Participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) and were deemed to be benefitting clinically despite progression, received a second course of pembrolizumab at the investigator's discretion. Pembrolizumab was administered at 200 mg IV on Day 1 of each 21-day cycle for up to 17 cycles (up to ~1 year additional).
- Placebo Switched Over to Pembrolizumab (Second Course): Participants who switched from saline placebo to complete the first course of up to 35 administrations of pembrolizumab (~2 years), initiated a second course of pembrolizumab at investigator's discretion. Pembrolizumab was administered 200 mg IV on Day 1 of each 21-day cycle for up to 17 cycles (up to ~1 year).
Arm/Group | Pembrolizumab + Chemotherapy Combo | Placebo + Chemotherapy | Placebo Switched Over to Pembrolizumab | Pembrolizumab Combo (Second Course) | Placebo Switched Over to Pembrolizumab (Second Course)
All-Cause Mortality (participants affected / at risk) | 225/278 | 143/281 | 111/118 | 6/12 | 0/1
Serious Adverse Events (participants affected / at risk) | 128/278 | 114/280 | 35/118 | 2/12 | 0/1
Other Adverse Events (participants affected / at risk) | 270/278 | 272/280 | 90/118 | 9/12 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy Combo (N=278) | Placebo + Chemotherapy (N=280) | Placebo Switched Over to Pembrolizumab (N=118) | Pembrolizumab Combo (Second Course) (N=12) | Placebo Switched Over to Pembrolizumab (Second Course) (N=1)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (15) | 10 (12) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (8) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (7) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 6 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 22 (23) | 21 (23) | 7 (9) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis migrans (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Chemotherapy Combo (N=278) | Placebo + Chemotherapy (N=280) | Placebo Switched Over to Pembrolizumab (N=118) | Pembrolizumab Combo (Second Course) (N=12) | Placebo Switched Over to Pembrolizumab (Second Course) (N=1)
Anaemia (Blood and lymphatic system disorders) | 148 (200) | 139 (186) | 17 (26) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 20 (46) | 20 (40) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 99 (201) | 85 (166) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 81 (131) | 64 (95) | 4 (6) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 20 (22) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 33 (36) | 6 (7) | 5 (6) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 22 (24) | 17 (17) | 3 (4) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 70 (93) | 62 (74) | 12 (14) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 88 (141) | 65 (86) | 16 (22) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 10 (12) | 3 (3) | 6 (7) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 6 (7) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 101 (151) | 90 (136) | 12 (13) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 14 (17) | 15 (16) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 51 (71) | 30 (47) | 6 (8) | 0 (0) | 0 (0)
Asthenia (General disorders) | 62 (83) | 60 (72) | 8 (16) | 0 (0) | 0 (0)
Chest pain (General disorders) | 20 (21) | 24 (24) | 9 (10) | 0 (0) | 0 (0)
Fatigue (General disorders) | 67 (92) | 72 (102) | 15 (15) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 26 (27) | 22 (30) | 3 (4) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 39 (45) | 35 (41) | 5 (7) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 22 (25) | 11 (12) | 5 (5) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (27) | 7 (7) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 14 (16) | 16 (16) | 5 (6) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 20 (30) | 10 (13) | 4 (7) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 16 (17) | 8 (9) | 7 (7) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 23 (39) | 12 (12) | 5 (9) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 26 (40) | 16 (17) | 6 (8) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 12 (19) | 12 (12) | 4 (5) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (13) | 3 (6) | 3 (6) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 26 (37) | 15 (24) | 11 (20) | 1 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 24 (59) | 28 (60) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 25 (52) | 23 (42) | 1 (1) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 31 (33) | 24 (24) | 11 (12) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 32 (78) | 32 (61) | 0 (0) | 1 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 77 (120) | 82 (101) | 9 (11) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 8 (9) | 7 (8) | 8 (10) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (14) | 12 (13) | 5 (7) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 (21) | 12 (19) | 7 (8) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (13) | 18 (27) | 4 (5) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (31) | 19 (28) | 8 (13) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 24 (36) | 21 (27) | 4 (4) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 20 (28) | 13 (14) | 7 (8) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (9) | 11 (17) | 7 (9) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 (103) | 48 (61) | 10 (13) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (24) | 37 (38) | 7 (7) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 37 (47) | 34 (41) | 3 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (31) | 27 (36) | 4 (4) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 21 (25) | 20 (23) | 4 (5) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 24 (27) | 11 (11) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 25 (28) | 23 (27) | 4 (9) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 60 (69) | 48 (56) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 21 (22) | 16 (17) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 33 (34) | 37 (39) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 15 (17) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 31 (32) | 23 (24) | 5 (5) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 49 (55) | 56 (66) | 12 (13) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 (46) | 45 (49) | 15 (15) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 (32) | 19 (21) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 23 (24) | 25 (36) | 12 (14) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 14 (21) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 13 (15) | 8 (8) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 128 (129) | 105 (106) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (12) | 8 (8) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 51 (61) | 25 (29) | 15 (18) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 52 (62) | 32 (37) | 7 (7) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 18 (22) | 14 (15) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 12 (13) | 16 (19) | 4 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT02775435/Prot_SAP_001.pdf